CLINICAL TRIAL: NCT03301480
Title: Contraceptive/HIV Affecting Risk in Adolescents
Acronym: CHARA
Status: Terminated | Type: Observational
Why Stopped: An interim review of the data revealed that there was broad inter-participant variability.The study was stopped due to futility.
Sponsor: University of Pittsburgh (Other)
Collaborators: National Institutes of Health (NIH) (NIH)
Responsible Party: Principal Investigator, Katherine Bunge, Assistant Professor, University of Pittsburgh
Other Study IDs: PRO17050002
Record Dates: First submitted 2017-08-08; First posted 2017-10-04 (Actual); Last update posted 2019-02-07 (Actual); Status verified 2019-02

CONDITIONS: Contraception; Hiv
MeSH Terms: conditions — Acquired Immunodeficiency Syndrome

STUDY DESIGN:
Observational Model: Case-Control | Time Perspective: Cross-Sectional
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (6):
- No contraception/18-19 years old
- Use of ENG-I/18 - 19 years old
- LNG-IUS/18-19 years old
- No Contraception/ 25 - 45 years old
- Use of ENG-I/25 - 45 years old
- LNG-IUS/25-45 years old

SUMMARY:
This study will evaluate the impact of hormonal contraceptives on HIV risk associated with changes to the innate immunity in the female genital tract in a cross-sectional study. HIV risk will be evaluated by the capacity of cervical tissue to replicate HIV when challenged ex vivo and correlated to the number of CD4 T cells, DCs, and macrophages; the capacity of cervicovaginal fluid to inhibit HIV will be correlated to soluble mucosal mediators, and the vaginal microbiota. The lower genital tract samples will be collected from 120 adolescents aged 18-19 (40 using no hormonal contraception, 40 using ENG-I, 40 using LNG-IUS). For comparison, 90 adult women aged 25-45 will be equally distributed between the same groupings.

ELIGIBILITY:
Inclusion Criteria:

1. Meets one of the following age groups (at the time of sample collection):

   1. Adolescent aged 18-19
   2. Adult aged 25-45
2. Meets one of the following contraception groups:

   1. Regular menstrual cycles by participant history (if not using hormonal contraception)
   2. Use of ENG-I (i.e. Implanon/Nexplanon) for at least 30 days by participant history
   3. Use of LNG-IUS (Mirena or Skyla) for at least 30 days by participant history
3. HIV uninfected Note: HIV testing will be done as part of screening. However, if a woman participated in a recent research study and has an HIV test result available from that study, this will suffice provided the date of the test is within 6 months of the study visit.
4. Willing to undergo pelvic exam and collection of cervical biopsies
5. Willing to provided written informed consent
6. Agree to be sexually abstinent for 48 hours prior to the cervical biopsies and for one week after the biopsies.

Exclusion Criteria:

1. Use of any other hormonal contraception other than ENG-I or LNG-IUS
2. Use of a diaphragm or spermicide for contraception
3. Pregnant or pregnancy within 90 days
4. Currently breastfeeding
5. Currently menstruating/bleeding (at time of specimen collection) Note: participant can return after cessation of bleeding for specimen collection
6. Past participation in more than one study involving cervical biopsies per participant report
7. Cervical biopsies within one month of specimen collection visit
8. Abnormal vaginal discharge or other genital tract symptoms at the time of specimen collection
9. Pelvic findings on the day of specimen collection consistent with cervicitis (i.e. MPC, erythema, edema) or anatomy making cervical biopsies difficult
10. Menopausal
11. Hysterectomy
12. History of malignancy of the genital tract (including cervix, uterus, vagina, and vulva)
13. History of immunosuppression (including HIV infection, diabetes, and chronic steroid use)
14. Known history of a platelet/bleeding/clotting disorder
15. Use of a systemic or vaginal antimicrobial agent within 7 days of specimen collection
16. Use of any vaginal product (i.e. douching, spermicide, lubricant) or device within 7 days of specimen collection Note: tampon use is acceptable
17. Any other condition that in the opinion of the Study Investigator would preclude provision of informed consent or make study participation unsafe, complicate the interpretation of study outcome data, or otherwise interfere with achieving the study objectives.

Ages: 18 Years to 45 Years | Sex: Female
Age Groups: Adult
Gender Based: Yes — participants must have a cervix for participation
Study Population: non-pregnant, HIV negative, healthy 18-19 year old women and 25-45 year old women
Sampling Method: Non-Probability Sample
Enrollment: 120 (Actual)
Dates: Start 2017-07-31 (Actual); Primary Completion 2018-09-17 (Actual); Study Completion 2018-09-17 (Actual)

PRIMARY OUTCOMES:
HIV replication in cervical tissue as measured by levels of HIV p24/viral transcripts | baseline
  cervical tissue testing
number of immune cells in cervical tissue, including CD45, CD3, CD4, and CD8 and their expression of CCR5, CCR6 and CD69, and CD11c+ DCs and CD14+ macrophages | baseline
  cervical tissue testing

SECONDARY OUTCOMES:
Prevalence of bacterial vaginosis defined as a Nugent score ≥7 on a vaginal smear | baseline
  vaginal specimen
prevalence and quantity of lactobacillus species and bacterial vaginosis associated bacteria as measured by traditional culture methods and quantitative PCR | baseline
  vaginal specimen
HIV inhibitory activity in mucosal fluid; and soluble mucosal factors identified through pathway analyses and confirmed by targeted ELISA/multiplexing technology (proteases/ anti-proteases, keratin, IFNε, and other molecules) | baseline
  mucosal fluid

CONTACTS AND LOCATIONS:
Overall Officials: Katherine Bunge, MD, Principal Investigator — University of Pittsburgh
Locations (1):
- Magee-Womens Hospital of UPMC, Pittsburgh, Pennsylvania, United States